CLINICAL TRIAL: NCT07015385
Title: Evaluation of a Novel Lip Bumper With Integrated Distal Shoe Appliance in Preventing Second Molar Impaction in Children With Anterior Deep Bite
Acronym: Novel Lip Bump
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dar Al Uloom University (Other)
Responsible Party: Principal Investigator, Sally Abd-ElMeniem ElHaddad, Assist. Prof., Dar Al Uloom University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33-06-2025
Record Dates: First submitted 2025-05-30; First posted 2025-06-11 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Bite; Orthodontics
Keywords: Malocclusion; Angle Class II; Deep Bite; Child
MeSH Terms: conditions — Bites and Stings; Malocclusion; Malocclusion, Angle Class II; Overbite

STUDY DESIGN:
Intervention Model Description: Parallel Assignment This clinical trial will follow a parallel assignment model, meaning participants will be randomly assigned to one of two independent groups, and each group will receive a distinct intervention throughout the duration of the study. There will be no crossover between groups.
  Group Assignments:
  Group I (Experimental Group):
  Participants will receive a lip bumper integrated with a distal shoe. This novel appliance aims to maintain space for the second molars and guide their eruption while simultaneously addressing anterior deep bite.
  Group II (Control Group):
  Participants will receive a conventional lip bumper, the standard interceptive appliance used to relieve lip pressure and promote arch development without specific design elements to prevent molar impaction.
  Key Characteristics of the Study Model:
  Allocation: Randomized Intervention Duration: 12 months
  Follow-Up Visits: Every 6 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lip Bumper with Integrated Distal Shoe (Experimental): Participants in this group will receive a novel orthodontic appliance that combines a traditional lip bumper with an integrated distal shoe. The appliance is designed to prevent mesial migration of the first molars and guide proper eruption of the second permanent molars. It also functions to relieve anterior deep bite by reducing lip pressure and promoting vertical and sagittal arch development. The appliance will be worn continuously for a period of 12 months with follow-up visits every 6 weeks for adjustments and monitoring.
  Interventions: Device: Lip Bumper with Integrated Distal Shoe
- Conventional Lip Bumper (Active Comparator): Participants in this group will receive a standard lip bumper appliance, commonly used in interceptive orthodontics to relieve lower arch crowding and eliminate lip pressure. This appliance does not include any mechanism to prevent mesial drift of the first molars or guide the eruption path of second molars. It will be used in the same time frame and follow-up schedule as the experimental group to allow direct comparison of outcomes.
  Interventions: Device: Conventional Lip Bumper

INTERVENTIONS:
Device: Lip Bumper with Integrated Distal Shoe — This novel appliance integrates a traditional lip bumper with a distal shoe extension designed to engage the mesial surface of the unerupted second permanent molar. The goal is to prevent mesial movement of the first molars and guide proper eruption of the second molars while simultaneously addressing anterior deep bite by eliminating lip pressure and promoting vertical incisor development. The device will be custom-fabricated for each participant and will be worn for 12 months, with clinical and radiographic evaluations conducted every 6 weeks.
  Arms: Lip Bumper with Integrated Distal Shoe
Device: Conventional Lip Bumper — The conventional lip bumper is an interceptive orthodontic appliance used to alleviate lower anterior crowding, eliminate perioral muscle pressure, and promote dental arch expansion. It does not include a distal shoe component and therefore offers no guidance for second molar eruption. This device will also be custom-fabricated and worn for 12 months, with scheduled monitoring every 6 weeks to assess treatment progress and compare outcomes with the experimental device.
  Arms: Conventional Lip Bumper

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a novel lip bumper with an integrated distal shoe in preventing second molar impaction in children aged 8-10 years with anterior open bite during the mixed dentition stage.

The main questions it aims to answer are:

* Does the integrated distal shoe significantly reduce the risk of second molar impaction compared to conventional lip bumpers?
* Does the appliance improve anterior open bite correction and influence lower incisor inclination?

Researchers will compare Group I (lip bumper with distal shoe) to Group II (conventional lip bumper) to see if the modified appliance prevents mesial drift of first molars and improves eruption outcomes of second molars.

Participants will:

* Undergo initial records including panoramic and cephalometric radiographs, study models, and intraoral photos
* Be fitted with one of the two appliances and followed up every 6 weeks over a 12-month period
* Receive radiographic and clinical evaluation of second molar eruption
* Complete assessments related to overbite changes, incisor inclination, comfort, and compliance This trial seeks to inform early orthodontic protocols and may offer a dual-function solution for both molar guidance and open bite correction.

DETAILED DESCRIPTION:
This clinical research study is focused on improving early orthodontic care for children who have an anterior deep bite-a condition where the upper teeth excessively overlap the lower front teeth-and are at risk of second molar impaction, a complication where the posterior teeth do not emerge properly. Left untreated, these issues can lead to long-term dental problems including poor bite alignment, crowding, or the need for surgical intervention.

Orthodontists often use a device called a lip bumper to reduce pressure from the lips on the lower front teeth, making room for crowded teeth and promoting healthy jaw development. However, a well-known downside of using a lip bumper-especially in young children-is that it can cause the first molars to drift forward. This forward movement can block the path for the second molars, increasing the risk that they will not erupt normally.

This study introduces a novel orthodontic appliance that aims to solve both problems at once. The new device combines the benefits of a traditional lip bumper with a "distal shoe"-a small guiding component that helps maintain proper space for the second molars to erupt. By doing so, it seeks not only to correct deep bite problems but also to prevent the common and serious issue of molar impaction.

The study will involve children between the ages of 8 and 10, a key stage of dental development. Participants will receive either the new dual-purpose device or a standard lip bumper and will be monitored over the course of a year. Throughout this period, researchers will examine how the teeth are moving, whether the posterior molars are erupting properly, and how well the deep bite is improving.

In addition to clinical evaluations, the study will gather feedback from children and their parents about comfort, ease of use, and any issues related to the appliance. Understanding patient experience is a vital part of assessing whether this new approach can be widely recommended in pediatric dental care.

Ultimately, this research aims to offer a more comprehensive and preventive solution for young patients undergoing early orthodontic treatment. If the new appliance proves effective, it could significantly reduce the need for more complex procedures later in life and promote better long-term dental health.

Ethical safeguards, including informed consent from parents and assent from participating children, are in place to ensure safety and understanding. The study has received institutional ethics approval and will be conducted under regular clinical monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 and 11 years
* In mixed dentition stage (presence of permanent first molars and incisors; unerupted second molars)
* Presence of an anterior deep bite of ≥ 2 mm (measured vertically between upper and lower incisors)
* Class I or mild Class II malocclusion
* Good general health with no systemic conditions that may affect dental development or treatment
* Written informed consent obtained from the parent or legal guardian and assent from the child

Exclusion Criteria:

* History of previous orthodontic treatment
* Presence of craniofacial anomalies (e.g., cleft lip/palate) or syndromic conditions
* Diagnosis of systemic diseases that affect bone metabolism or craniofacial growth (e.g., juvenile rheumatoid arthritis, osteogenesis imperfecta)
* Evidence of poor oral hygiene or active caries requiring urgent dental care
* Use of any medication known to affect dental development (e.g., long-term corticosteroids, antiepileptics)
* Behavioral or developmental disorders that would preclude cooperation with appliance wear or study procedures

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Radiographic Assessment of Second Molar Eruption Angle and Position | At baseline and after 12 months of appliance use
  Radiographic Eruption Angle Measurement Scale (in degrees)
  Objectives:
  To evaluate the effect of the appliance on the eruption trajectory and final position of the second permanent molars, using radiographic measurements to detect impaction or favorable eruption patterns.
  * Measurement Method: Panoramic radiograph using digital angle analysis tools to measure the angle between the long axis of the second molar and a stable reference line (e.g., occlusal plane or mandibular base).
  * Scale Range:
    * Minimum value: 0° (perfect vertical eruption)
    * Maximum value: ~90° (severely impacted or horizontal position)
  * Interpretation:
    * Lower scores (closer to 0°) indicate a more favorable eruption position and vertical alignment.
    * Higher scores (closer to 90°) indicate a worse outcome, suggesting impaction or abnormal angulation.
  Angular and positional changes of the mandibular second permanent molars (in degrees or millimeters) as observed on standardized panoramic radiographs

SECONDARY OUTCOMES:
Change in Overbite (in mm) | Baseline and 12 months
  Measurement Method: Measured on study models from the incisal edge of the maxillary central incisor to the incisal edge of the opposing mandibular incisor at the point of greatest overlap, when posterior teeth are in occlusion.
  Scale Range:
  Minimum value: 0 mm (edge-to-edge or open bite)
  Maximum value: Typically up to 6-8 mm (deep bite), depending on the patient's anatomy
  Interpretation:
  Lower scores after treatment indicate improvement (reduced deep bite), representing a better clinical outcome Higher scores after treatment suggest persistence or worsening of the deep bite, representing a worse clinical outcome
Lower Incisor Inclination (IMPA - Incisor Mandibular Plane Angle) in degrees | Baseline and 12 months
  Measurement Method:
  IMPA is measured on standardized lateral cephalometric radiographs as the angle between the long axis of the most prominent mandibular central incisor and the mandibular plane (typically drawn from gonion to menton).
  Scale Range:
  Minimum value: ~80° (retroclined lower incisors) Maximum value: ~110° (proclined lower incisors) (Typical normal range: 90° ± 5°)
  Interpretation:
  Lower scores (e.g., < 85°) indicate retroclination of the lower incisors Higher scores (e.g., > 95°) indicate proclination
Visual Analog Scale for Orthodontic Comfort and Tolerance (0-10 scale) Patient-Reported Comfort and Appliance Tolerance | 1 week, 6 weeks, 3 months, and 12 months
  Patients will complete a self-reported questionnaire at specified intervals (1 week, 6 weeks, 3 months, and 12 months) rating their comfort and tolerance of the appliance. The scale used is a Visual Analog Scale (VAS) ranging from 0 to 10.
  Scale Range:
  Maximum value: 10 = No comfort at all / appliance is very uncomfortable and intolerable Minimum value: 0 = Very comfortable / appliance is completely tolerable
  Interpretation:
  Lower scores indicate better outcomes, reflecting greater comfort and tolerance to the appliance
  Higher scores suggest discomfort, poor adaptation, or potential complications impacting patient compliance
Orthodontic Appliance Compliance Assessment Scale (0-5 scale) | at each follow-up visit (every 6 weeks)
  Orthodontist will assess patient compliance based on appliance wear, cleanliness, and adherence to instructions. Scoring will be based on clinical observation and patient self-report, using a standardized 6-point scale.
  Scale Range:
  0: Non-compliant - never wears appliance or refuses treatment
  1. Very poor compliance - wears appliance <25% of the time
  2. Poor compliance - inconsistent use, visible neglect of hygiene
  3. Moderate compliance - wears appliance ~50-75% of expected time
  4. Good compliance - minor lapses in wear or cleaning
  5. Excellent compliance - wears appliance as instructed, maintains hygiene
  Interpretation:
  Higher scores (4-5) reflect better outcomes, indicating strong adherence to treatment and greater likelihood of therapeutic success
  Lower scores (0-2) indicate poor cooperation, which may reduce treatment effectiveness
Soft Tissue Reaction Severity Scale (0-3 score per site) | At each 6-week follow-up visit
  Clinical examination will be performed to assess the soft tissues adjacent to the appliance. Adverse reactions such as ulceration, erythema, swelling, and hyperplasia will be documented using a standardized 4-point severity scale.
  Scale Range:
  0: No reaction - healthy tissue
  1. Mild - slight redness or irritation, no ulceration
  2. Moderate - noticeable inflammation, small ulcers or discomfort
  3. Severe - pronounced ulceration, swelling, or tissue overgrowth requiring intervention
  Interpretation:
  Lower scores (0-1) indicate better outcomes, reflecting good appliance biocompatibility and patient adaptation Higher scores (2-3) indicate worse outcomes, signifying poor tissue response or intolerance to the appliance

IPD SHARING:
Plan to Share IPD: Yes
The following de-identified individual participant data (IPD) will be shared:
  Demographic data: age, sex, and baseline dental classification (e.g., type of malocclusion)
  Radiographic measurements: second molar eruption angle and position at baseline and 12 months
  Cephalometric data: baseline and post-treatment incisor mandibular plane angle (IMPA)
  Overbite measurements: baseline and post-treatment vertical overlap (in mm)
  Patient-reported outcomes: responses from comfort and compliance questionnaires
  Adverse event reports: type, frequency, and severity of any soft tissue complications
  Compliance assessments: clinician-rated appliance wear and follow-up adherence
  All shared data will be fully anonymized in accordance with ethical standards and privacy regulations.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD Availability Timeline
  Start Date for IPD Availability:
  Six months after publication of the primary study results in a peer-reviewed journal.
  End Date for IPD Availability:
  Five years from the start date of data sharing.
  During this period, de-identified individual participant data and related supporting documents (such as the study protocol and statistical analysis plan) will be made available to qualified researchers upon reasonable request and subject to data use agreements.